CLINICAL TRIAL: NCT02348281
Title: A Prospective, Single Center, Phase II Study of Bicalutamide as A Treatment in Androgen Receptor (AR)-Positive Metastatic Triple-Negative Breast Cancer (mTNBC) Patients
Brief Title: Bicalutamide as A Treatment in AR-positive Metastatic Triple-Negative Breast Cancer (mTNBC) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: it's too slow to enroll suitable patients into this study
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, M.D.,Ph.D., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2015-17
Record Dates: First submitted 2015-01-18; First posted 2015-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: triple negative breast cancer; androgen receptor; bicalutamide
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bicalutamide (Experimental): 150mg, po, qd, d1-28
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide — 150mg, po, qd, d1-28
  Other Names: Casodex

SUMMARY:
This prospective, single center, phase II study is to evaluate the efficacy and safety of bicalutamide as a treatment in androgen receptor (AR)-positive metastatic triple-negative breast cancer (mTNBC) patients.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is defined as the absence of estrogen and progesterone receptor expression as well as ERBB2 amplification. It has no response to endocrine or anti-ERBB2 therapies. Recent studies have found some potential therapeutic targets for TNBC. However, it still has a poor outcome. It was reported that TNBC has six subtypes, including 2 basal-like (BL1 and BL2), an immunomodulatory (IM), a mesenchymal (M), a mesenchymal stem-like (MSL), and a luminal androgen receptor (LAR) subtype. Different subtype may be sensitive to different treatment. Bicalutamide is an oral, non-steroidal, androgen receptor (AR) antagonist. It is approved by the Food and Drug Administration (FDA) for the treatment of metastatic prostate cancer. Recently, a study explored the efficacy of bicalutamide in AR positive, estrogen receptor negative metastatic breast cancer (MBC), which showed a high clinical benefit rate (CBR) and a good safety profile. Based on the above reasons, we initiate this phase II study to evaluate the efficacy and safety of bicalutamide in AR positive metastatic triple-negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Females elder than 18
2. Histological proven unresectable or metastatic breast cancer patients who underwent at least one chemotherapy regimen for metastatic disease
3. Patients with androgen Receptor (AR) positive (IHC >10% nuclear staining) either for primary tumor or metastatic lesion
4. Triple-negative for estrogen receptor (ER), progestogen receptor (PR), and human epithelial receptor-2 (HER2) by IHC (ER <1%, PR <1% and Her2 negative). A negative Her2 gene amplification should be verified by FISH test for those patients with Her2 (2+). For those with Her2 (1+), FISH test might be considered by the investigator.
5. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1)
6. Performance status no more than 2
7. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
8. Life expectancy longer than 12 weeks
9. No serious medical history of heart, lung, liver and kidney
10. Be able to understand the study procedures and sign informed consent.
11. Patients with good compliance

Exclusion Criteria:

1. Pregnant or lactating women
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study
3. Patients treated with an investigational product within 4 weeks before the enrollment
4. Patients who received chemotherapy within 4 weeks before the enrollment
5. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
6. Other active malignancies (including other hematologic malignancies) or other malignancies within the last 5 years, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
7. Patients having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
8. Uncontrolled serious infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | every 8 weeks, up to 48 weeks
  Clinical benefit rate is defined as the percentage of patients who achieve complete response (CR), partial response (PR) and stable disease (SD) ≥24 weeks by RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) | every 8 weeks, up to 24 weeks
  Objective response rate is defined as the percentage of patients who achieve complete response (CR) and partial response (PR) by RECIST version 1.1 criteria.
Progression free survival (PFS) | every 8 weeks, up to 48 months
  Progression free survival is defined as the time from enrollment to the first documented disease progression or death from any cause.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | every 4 weeks, up to 24 weeks
  Evaluate incidence of adverse events and severity grade of these events
Overall Survival (OS) | every 3 months, up to 100 months
  Overall Survival is defined as the time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, M.D., Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China